CLINICAL TRIAL: NCT04681677
Title: Phase II Study of Patients With Recurrent Glioblastoma Multiforme Treated With Maximal Safe Neurosurgical Resection and Intra-Operative Radiation Therapy (IORT) Using the Xoft Axxent Electronic Brachytherapy System and Bevacizumab
Brief Title: Recurrent GBM Treated With Neurosurgical Resection and IORT Using the Xoft Axxent eBx System and Bevacizumab
Acronym: IORT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unspecified business decision
Sponsor: Xoft, Inc. (Industry)
Collaborators: Icad, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTPR-0017
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; GBM; Recurrent GBM
Keywords: Bevacizumab; Glioblastoma; Recurrent Glioblastoma; GBM; Recurrent GBM; IORT; Intra-Operative Radiation Therapy; Avastin
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Single arm, prospective, multi-center, non-randomized, historical control, non-inferiority study of subjects treated with single fraction, Intra-Operative Radiation Therapy at the time of maximal resection for recurrent GBM. Treatment with Bevacizumab will be initiated 28-56 days after surgery depending on surgical wound healing assessment at the discretion of the treating investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental: Intra-operative Radiation Therapy - IORT (Experimental): Radiation: Intra-operative Radiation Therapy - IORT
  Interventions: Radiation: Radiation: Intra-operative Radiation Therapy - IORT; Drug: Bevacizumab

INTERVENTIONS:
Radiation: Radiation: Intra-operative Radiation Therapy - IORT — Single fraction, Intra-operative Radiation Therapy at the time of surgical resection of recurrent GBM followed by Bevacizumab 28-56 days after surgery.
Drug: Bevacizumab — Bevacizumab
  Other Names: Avastin

SUMMARY:
The purpose of this trial is to assess the overall survival of patients treated with the Xoft Axxent eBx System and post-radiation adjuvant Bevacizumab for single-fraction IORT following maximal neurosurgical resection of recurrent glioblastoma. A historical comparison will be made to the results of the EBRT + Bevacizumab arm of RTOG 1205.

DETAILED DESCRIPTION:
The rationale for IORT, as the sole radiation therapy following surgical resection of recurrent GBM is to expand upon the favorable preliminary results in feasibility, safety and efficacy outcomes obtained at the European Medical Center Study Group (EMC Study Group). The rationale to add Bevacizumab as a systemic treatment is to target radio-resistant and highly tumorigenic cancer stem cells as well as to benefit from its radioprotective effects, i.e. reducing risk of radiation necrosis. Lastly, using Bevacizumab as a systemic therapy will enable the comparison of the results to the historic control arm, the EBRT arm of RTOG 1205.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has the ability to provide written informed consent
2. Subject has the willingness to comply with all study procedures for the duration of the study
3. Subject has histopathologically proven diagnosis of GBM or variants (gliosarcoma, giant cell glioblastoma etc.). Subjects will be also eligible if the original histology was lower-grade glioma and a subsequent diagnosis of glioblastoma or gliosarcoma is made.
4. Subjects must have shown unequivocal radiographic evidence for tumor progression by contrast-enhanced MRI within 21 days prior to enrollment
5. Subjects must have passed an interval of 6 months or greater between completion of prior radiotherapy and enrollment. If subjects have not passed an interval of at least 6 months, they may still be eligible if they meet one or more of the following criteria:

   1. New areas of tumor outside the original radiotherapy fields as determined by the investigator, or
   2. Histologic confirmation of tumor through biopsy or resection, or
   3. Nuclear medicine imaging, MR spectroscopy, or MR perfusion imaging consistent with true progressive disease, rather than radiation necrosis obtained within 28 days of registration AND an interval of at least 90 days between completion of radiotherapy and enrollment
6. The recurrent GBM must be potentially-resectable with the intent to resect such that residual tumor rim is less than 1 cm enhancing disease
7. The recurrent GBM must have the appropriate dimensions to allow a Xoft applicator balloon to fit into the tumor cavity
8. Subject has prior history of standard dose CNS radiation of 60 Gy in 30 fractions or 59.4 Gy in 1.8 Gy fractions, or equivalent of lower doses. Patients who have received prior treatment with non-standard RT dose and fractionation, interstitial brachytherapy, stereotactic radiosurgery, etc. are eligible as long as the criterion in 5. is met or approved by principal investigator.
9. Subjects who have undergone CNS related core or needle biopsies, a minimum of 7 days must have elapsed prior to registration
10. History/physical examination, including neurologic examination, within 14 days prior to enrollment (i.e. date the informed consent was signed by the patient)
11. Subject must be ≥ 18 years of age
12. Subject must have a Karnofsky Performance Score ≥ 60%
13. Subject will have had a CBC/differential obtained within 14 days prior to enrollment , with adequate bone marrow function, i.e.:

    d) Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3 e) Platelets ≥ 75,000 cells/mm3 f) Hemoglobin ≥ 9.0 g/dl (The use of transfusion or other intervention to achieve Hgb ≥ 9.0 g/dl is acceptable.)
14. Subjects liver and renal function test should reflect adequate hepatic and renal function 14 days prior to enrollment, i.e.:

    1. Total bilirubin ≤ 2.0 mg/dL, and SGOT or AST ≤ 2.5 times the upper limit of normal
    2. Serum creatinine ≤ 1.8 mg/dL) within 14 days prior to enrollment
15. Subject urine protein level must reflect the following requirements within 14 days before enrollment:

    1. Urine protein: creatinine (UPC ) ratio < 1.0 OR
    2. Urine dipstick for proteinuria ≤ 2+ (patients who have > 2+ proteinuria on dipstick urinalysis at baseline, must have an UPC ratio <1.0 to be eligible. If the UPC ratio is ≥ 1.0, subsequent 24 hrs urine collection must be ≤ 1 g protein in 24 hrs)
16. Patients on full-dose anticoagulants (e.g., warfarin or LMW heparin) must meet both of the following criteria:

    1. No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices).
    2. In-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin, within 14 days prior to enrollment.
17. Women of child-bearing potential must have a negative pregnancy test within 7 days of treatment
18. Subjects of child-bearing potential must agree to use adequate contraceptive precautions and not to breastfeed (if applicable) until six months after the end of the treatment with Bevacizumab.
19. Patient is planned to have surgery for recurrent Glioblastoma

Exclusion Criteria:

1. Subject has had more than three relapses
2. Subject has multi-centric disease
3. Subject has tumors in or near (less than 10mm from tumor margin) critical brain structures, that would exclude sufficient dose delivery to the tumor margin:

   1. Optic Chiasm
   2. Optic Nerve
4. Subject has infratentorial, or leptomeningeal evidence of recurrent disease
5. Subject has recurrent or persistent tumor greater than 6 cm in maximum diameter
6. Subject underwent prior therapy with an inhibitor of VEGF or VEGFR (including Bevacizumab)
7. Subject suffered from prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1 year (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
8. Women who are pregnant or nursing. Women with child-bearing potential or sexually active men that are not willing/able to use medically acceptable forms of contraception.
9. Subject has contraindications for MRI with or without gadolinium.
10. Subject has contraindications for anesthesia or surgery.
11. Subject is on another therapeutic clinical trial concurrently.
12. Subject suffers severe, active co-morbidity, defined as follows:

    1. Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to enrollment
    2. Transmural myocardial infarction within the last 6 months prior to enrollment
    3. History of stroke or transient ischemic attack within 6 months prior to enrollment
    4. Significant vascular (aortic) disease or clinically significant peripheral vascular disease
    5. Active venous or arterial thromboembolic disease
    6. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of enrollment
    7. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of enrollment
    8. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects. Laboratory tests for liver function other than screening panel coagulation parameters are not required for entry into this protocol
    9. Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition. HIV testing is not required for entry into this protocol.
13. Prior history of hypertensive crisis or hypertensive encephalopathy
14. Subject has history of a non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to enrollment
15. Subject suffers from gastrointestinal bleeding or any other hemorrhage /bleeding event CTCAE v.5 grade 3 or greater within 30 days prior to enrollment
16. Subject suffers from Hypersensitivity to Bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
median overall survival (mOS) | 3 Years
  The median overall survival (mOS) of subjects treated with the Xoft Axxent Electronic Brachytherapy (eBx)® System when used for single-fraction, intra-operative radiation therapy (IORT) following maximal safe neurosurgical resection of recurrent glioblastoma and bevacizumab and compare it to the EBRT + Bevacizumab arm of RTOG 1205.

SECONDARY OUTCOMES:
6 Month rate progression-free survival (PFS) | 6 Month
  To assess progression-free survival and compare it to the EBRT + Bevacizumab arm of RTOG 1205.
tumor progression at four weeks | 4 Weeks
  To assess the tumor progression in the first four weeks after surgery
Local and distant progression-free survival | 3 Years
  To assess local and distant progression free survival
Quality of Life and radiation-related neurotoxicity | 3 Years
  To assess Quality of Life (QOL) and radiation-related neurotoxicity and compare it to the EBRT + Bevacizumab arm of RTOG 1205.
Rate of adverse events/safety | 3 Years
  To assess the rate of adverse events/ safety and compare it to the EBRT + Bevacizumab arm of RTOG 1205

OTHER OUTCOMES:
imaging changes | 3 Years
  To characterize the pattern of failure based on a centralized MRI review

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- Providence Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Background] Louis DN, Perry A, Reifenberger G, von Deimling A, Figarella-Branger D, Cavenee WK, Ohgaki H, Wiestler OD, Kleihues P, Ellison DW. The 2016 World Health Organization Classification of Tumors of the Central Nervous System: a summary. Acta Neuropathol. 2016 Jun;131(6):803-20. doi: 10.1007/s00401-016-1545-1. Epub 2016 May 9. PMID 27157931
- [Background] Stupp R, Tonn JC, Brada M, Pentheroudakis G; ESMO Guidelines Working Group. High-grade malignant glioma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2010 May;21 Suppl 5:v190-3. doi: 10.1093/annonc/mdq187. No abstract available. PMID 20555079
- [Background] Goryaynov SA, Gol'dberg MF, Golanov AV, Zolotova SV, Shishkina LV, Ryzhova MV, Pitskhelauri DI, Zhukov VY, Usachev DY, Belyaev AY, Kondrashov AV, Shurkhay VA, Potapov AA. [The phenomenon of long-term survival in glioblastoma patients. Part I: the role of clinical and demographic factors and an IDH1 mutation (R 132 H)]. Zh Vopr Neirokhir Im N N Burdenko. 2017;81(3):5-16. doi: 10.17116/neiro20178135-16. Russian. PMID 28665384
- [Background] Haj A, Doenitz C, Schebesch KM, Ehrensberger D, Hau P, Putnik K, Riemenschneider MJ, Wendl C, Gerken M, Pukrop T, Brawanski A, Proescholdt MA. Extent of Resection in Newly Diagnosed Glioblastoma: Impact of a Specialized Neuro-Oncology Care Center. Brain Sci. 2017 Dec 25;8(1):5. doi: 10.3390/brainsci8010005. PMID 29295569
- [Background] Hardesty DA, Sanai N. The value of glioma extent of resection in the modern neurosurgical era. Front Neurol. 2012 Oct 18;3:140. doi: 10.3389/fneur.2012.00140. eCollection 2012. PMID 23087667
- [Background] Krivoshapkin AL, Sergeev GS, Gaytan AS, Kurbatov VP, Kalneus LE, Tarantsev EG. New software for objective evaluation of brain glioblastoma resection degree. Zh Vopr Neirokhir Im N N Burdenko. 2014;78(5):33-9; discussion 40. English, Russian. PMID 25406906
- [Background] Davis ME. Glioblastoma: Overview of Disease and Treatment. Clin J Oncol Nurs. 2016 Oct 1;20(5 Suppl):S2-8. doi: 10.1188/16.CJON.S1.2-8. PMID 27668386
- [Background] Gaspar LE, Fisher BJ, Macdonald DR, LeBer DV, Halperin EC, Schold SC Jr, Cairncross JG. Supratentorial malignant glioma: patterns of recurrence and implications for external beam local treatment. Int J Radiat Oncol Biol Phys. 1992;24(1):55-7. doi: 10.1016/0360-3016(92)91021-e. PMID 1512163
- [Background] Choucair AK, Levin VA, Gutin PH, Davis RL, Silver P, Edwards MS, Wilson CB. Development of multiple lesions during radiation therapy and chemotherapy in patients with gliomas. J Neurosurg. 1986 Nov;65(5):654-8. doi: 10.3171/jns.1986.65.5.0654. PMID 3021931
- [Background] Mallick S, Benson R, Hakim A, Rath GK. Management of glioblastoma after recurrence: A changing paradigm. J Egypt Natl Canc Inst. 2016 Dec;28(4):199-210. doi: 10.1016/j.jnci.2016.07.001. Epub 2016 Jul 28. PMID 27476474
- [Background] Weller M, van den Bent M, Tonn JC, Stupp R, Preusser M, Cohen-Jonathan-Moyal E, Henriksson R, Le Rhun E, Balana C, Chinot O, Bendszus M, Reijneveld JC, Dhermain F, French P, Marosi C, Watts C, Oberg I, Pilkington G, Baumert BG, Taphoorn MJB, Hegi M, Westphal M, Reifenberger G, Soffietti R, Wick W; European Association for Neuro-Oncology (EANO) Task Force on Gliomas. European Association for Neuro-Oncology (EANO) guideline on the diagnosis and treatment of adult astrocytic and oligodendroglial gliomas. Lancet Oncol. 2017 Jun;18(6):e315-e329. doi: 10.1016/S1470-2045(17)30194-8. Epub 2017 May 5. PMID 28483413
- [Background] van Linde ME, Brahm CG, de Witt Hamer PC, Reijneveld JC, Bruynzeel AME, Vandertop WP, van de Ven PM, Wagemakers M, van der Weide HL, Enting RH, Walenkamp AME, Verheul HMW. Treatment outcome of patients with recurrent glioblastoma multiforme: a retrospective multicenter analysis. J Neurooncol. 2017 Oct;135(1):183-192. doi: 10.1007/s11060-017-2564-z. Epub 2017 Jul 20. PMID 28730289
- [Background] Ringel F, Pape H, Sabel M, Krex D, Bock HC, Misch M, Weyerbrock A, Westermaier T, Senft C, Schucht P, Meyer B, Simon M; SN1 study group. Clinical benefit from resection of recurrent glioblastomas: results of a multicenter study including 503 patients with recurrent glioblastomas undergoing surgical resection. Neuro Oncol. 2016 Jan;18(1):96-104. doi: 10.1093/neuonc/nov145. Epub 2015 Aug 4. PMID 26243790
- [Background] Landy HJ, Feun L, Schwade JG, Snodgrass S, Lu Y, Gutman F. Retreatment of intracranial gliomas. South Med J. 1994 Feb;87(2):211-4. doi: 10.1097/00007611-199402000-00013. PMID 8115886
- [Background] Ammirati M, Galicich JH, Arbit E, Liao Y. Reoperation in the treatment of recurrent intracranial malignant gliomas. Neurosurgery. 1987 Nov;21(5):607-14. doi: 10.1227/00006123-198711000-00001. PMID 2827051
- [Background] Harsh GR 4th, Levin VA, Gutin PH, Seager M, Silver P, Wilson CB. Reoperation for recurrent glioblastoma and anaplastic astrocytoma. Neurosurgery. 1987 Nov;21(5):615-21. doi: 10.1227/00006123-198711000-00002. PMID 2827052
- [Background] Pace A, Dirven L, Koekkoek JAF, Golla H, Fleming J, Ruda R, Marosi C, Le Rhun E, Grant R, Oliver K, Oberg I, Bulbeck HJ, Rooney AG, Henriksson R, Pasman HRW, Oberndorfer S, Weller M, Taphoorn MJB; European Association of Neuro-Oncology palliative care task force. European Association for Neuro-Oncology (EANO) guidelines for palliative care in adults with glioma. Lancet Oncol. 2017 Jun;18(6):e330-e340. doi: 10.1016/S1470-2045(17)30345-5. PMID 28593859
- [Background] Lederman G, Wronski M, Arbit E, Odaimi M, Wertheim S, Lombardi E, Wrzolek M. Treatment of recurrent glioblastoma multiforme using fractionated stereotactic radiosurgery and concurrent paclitaxel. Am J Clin Oncol. 2000 Apr;23(2):155-9. doi: 10.1097/00000421-200004000-00010. PMID 10776976
- [Background] Young B, Oldfield EH, Markesbery WR, Haack D, Tibbs PA, McCombs P, Chin HW, Maruyama Y, Meacham WF. Reoperation for glioblastoma. J Neurosurg. 1981 Dec;55(6):917-21. doi: 10.3171/jns.1981.55.6.0917. PMID 6271933
- [Background] Bloch O, Han SJ, Cha S, Sun MZ, Aghi MK, McDermott MW, Berger MS, Parsa AT. Impact of extent of resection for recurrent glioblastoma on overall survival: clinical article. J Neurosurg. 2012 Dec;117(6):1032-8. doi: 10.3171/2012.9.JNS12504. Epub 2012 Oct 5. PMID 23039151
- [Background] Ruben JD, Dally M, Bailey M, Smith R, McLean CA, Fedele P. Cerebral radiation necrosis: incidence, outcomes, and risk factors with emphasis on radiation parameters and chemotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):499-508. doi: 10.1016/j.ijrobp.2005.12.002. Epub 2006 Mar 6. PMID 16517093
- [Background] Zamzuri I, Rahman GI, Muzaimi M, Jafri AM, Nik Ruzman NI, Lutfi YA, Biswal BM, Nazaruddin HW, Mar W. Polymodal therapy for high grade gliomas: a case report of favourable outcomes following intraoperative radiation therapy. Med J Malaysia. 2012 Feb;67(1):121-2. PMID 22582564
- [Background] Scanderbeg DJ, Alksne JF, Lawson JD, Murphy KT. Novel use of the Contura for high dose rate cranial brachytherapy. Med Dosim. 2011 Winter;36(4):344-6. doi: 10.1016/j.meddos.2010.08.001. Epub 2010 Dec 8. PMID 21144735